CLINICAL TRIAL: NCT02370719
Title: Evaluation of an mHealth Behavioural Intervention for the Self-Management for Type 2 Diabetes Mellitus
Brief Title: Evaluation of an mHealth Behavioural Intervention for the Self-Management for Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the inability to recruit the required number of participants, the study has been terminated.
Sponsor: University Health Network, Toronto (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); University of Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joseph Cafazzo, Senior Director, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BantII
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; Randomized controlled trial; Primary care; Physical activity; Lifestyle; Blood glucose; Mobile health; Hb A1c; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Mobile application plus standard of care
  Interventions: Behavioral: Mobile application for diabetes self-management
- Control Group (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Mobile application for diabetes self-management
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to evaluate a patient-centered diabetes self-management mobile application (app), which was developed with feedback from both patients and healthcare providers. During the 12 month randomized control trial, participants in the intervention group will be provided with a mobile phone and commercial home medical devices, such as a weight scale, glucometer and activity monitor. The measurements taken from the medical devices will wirelessly transfer to the mobile phone, where the app will assess the data and provide patients with actionable self-management knowledge. The proposed intervention may be helpful in increasing adherence to recommended self-care practices, improving self-efficacy, and enhancing the overall patient experience.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking individuals
* Diagnosed with non-insulin requiring type 2 diabetes
* Outpatients
* Baseline A1c of 7.5% or higher

Exclusion Criteria:

* Patients who are deemed unable to use a mobile phone (e.g. due to vision problems), and/or to comply with home monitoring (e.g. suffering from anxiety or depression)
* Diabetes duration <1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06-28; Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to 12 months | Baseline, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Blood pressure | Baseline, 3, 6, 9 and 12 months
Weight | Baseline, 3, 6, 9 and 12 months
Cholesterol (LDL and total) | Baseline, 6 and 12 months
Medication changes | 3, 6, 9 and 12 months
Glycemic excursions | 3, 6, 9 and 12 months
BMI | Baseline, 3, 6, 9 and 12 months
Diabetes Distress Scale | Baseline, 6 and 12 months
Diabetes Empowerment Scale | Baseline, 6 and 12 months
Summary of Diabetes Self-Care Activities | Baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Cafazzo, PEng, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Goyal S, Lewis G, Yu C, Rotondi M, Seto E, Cafazzo JA. Evaluation of a Behavioral Mobile Phone App Intervention for the Self-Management of Type 2 Diabetes: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2016 Aug 19;5(3):e174. doi: 10.2196/resprot.5959. PMID 27542325